CLINICAL TRIAL: NCT03845322
Title: Clinical Action of Curcumin/Turmeric in Chronic Subdural Hematoma Recurrence
Brief Title: Curcumin/Turmeric as a Treatment for Patients With Subdural Hematomas Recurrence
Acronym: CACTIS
Status: Withdrawn | Phase: Early Phase 1 | Type: Interventional
Why Stopped: 12 Screen failures and Changes in PI and loss of residency program.
Sponsor: University of New Mexico (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 17-348
Record Dates: First submitted 2019-02-07; First posted 2019-02-19 (Actual); Last update posted 2022-05-25 (Actual); Status verified 2019-02

CONDITIONS: Hematoma, Subdural, Chronic
Keywords: curcumin; chronic; recurrence; hematoma; subdural; turmeric
MeSH Terms: conditions — Hematoma, Subdural, Chronic; Bronchiolitis Obliterans Syndrome; Recurrence; Hematoma | interventions — Curcumin

STUDY DESIGN:
Intervention Model Description: This is an experimental study, each consented subject will be instructed that he/she will be randomized to either the placebo group or the curcumin group.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: This is a double-blinded, randomized placebo-controlled pilot study. The patients, neurosurgeons, nurses and clinical coordinators will be blinded except for the research pharmacists who will keep a key linking a code # on a bottle handed to the clinical coordinator and the patient's medical record number (MRN #). The pill bottles handed to the clinical coordinator will be identical for placebo and CC.
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Curcumin pills group (Experimental): 24 Patient will receive Curcumin (CC) pills, within 24 hours post-operatively (as long as they are able to take oral medication). It will then be continued TID
  Interventions: Drug: Curcumin Pill
- Placebo group (Placebo Comparator): 24 Patient will receive Placebo pills, within 24 hours post-operatively (as long as they are able to take oral medication. It will then be continued TID.
  Interventions: Drug: Placebo pills

INTERVENTIONS:
Drug: Curcumin Pill — Curcumin (turmeric extract), over the counter supplement (1 capsule/three times a day). According to the Company, each capsule contains: 270 mg of pure curcuminoids (curcumin) and 3 mg of black pepper extract. Recommended serving size is 3 capsules per day in total, the patients will receive 810 mg of pure curcumin and 9 mg of black pepper extract (peperine/BioPerine) per day.
  Arms: Curcumin pills group
Drug: Placebo pills — The placebo pill is a vegetarian cellulose capsule, with cellulose powder inside. The composition is cellulose and magnesium stearate.
  Arms: Placebo group

SUMMARY:
Our long-term objective is to evaluate the efficacy of curcumin (CC) in preventing a recurrence of chronic subdural hematoma (cSDH) following surgical evacuation. Recurrence is defined as an increase in total hematoma volume on the operated side compared to a post-operative day one CT scan with persistent or recurrent neurological symptoms. The investigators propose this pilot study to assess feasibility and obtain preliminary benefit assessment of the proposed therapeutic approach.

Objective 1: To determine if the use of CC treatment reduces the total hematoma cavity volume over a 6-month interval, compared to a post-subdural drain removal CT scan. This evaluation is expected to offer sufficient evidence for a larger definitive trial.

Objective 2: Study the effect of CC on interleukin-8 (IL-8)-induced disruption of endothelial permeability in vitro using human vascular endothelial cells.

Central hypothesis: CC treatment prevents the re-accumulation of cSDH, which may occur by inhibition of IL-8 and allowing resolution of the total hematoma cavity volume over six months.

DETAILED DESCRIPTION:
Chronic subdural hematomas (cSDH) are extra-axial fluid collections in the cranium that can result in brain compression and neurological decline. cSDH commonly occurs after traumatic brain injury (TBI); though, many times there is no history of trauma. The incidence of cSDH is expected to significantly rise, due to an increasing elderly population worldwide.This is a common and challenging neurosurgical problem due to their ability to recur requiring repeated surgical reevacuation. Repeat surgery comes with additional morbidity as well as rising costs for both patients and hospitals. Operative decompression is the treatment of choice; however, an effective therapy preventing recurrence of cSDH after surgical intervention has not yet been found. Our long-term goal is to develop a therapeutic approach focused on the prevention of cSDH recurrence after initial surgical intervention.

The current literature and our own preliminary data have demonstrated that there is local elevation of pro-inflammatory chemokines and pro-angiogenic factors within the subdural hematoma cavity of chronic subdural hematomas that are not found systemically. Interleukin-8 (IL8 or chemokine (C-X-C motif) ligand 8, CXCL8) demonstrates both pro-inflammatory and pro-angiogenic properties. Curcumin has shown to directly inhibit the production and activity of CXCL-8 (IL-8) in vitro and in vivo, as well as down regulating the activity of VEGF (vascular endothelial growth factor) and bFGF (basic fibroblast growth factor). These combined effects make CC an important anti-inflammatory and antiangiogenic molecule that has the potential to reduce the recurrence rate of chronic subdural hematomas. The investigators expect that CC will prevent/reduce persistent hemorrhage within the subdural hematoma cavity, by blocking IL-8-induced disruption of the blood vessels. Specifically, CC is expected to preserve blood vessel leakage and accumulation of blood in SDH cavity, by blocking destructive effect of IL-8 on the vascular endothelial tight junctions.

CC has demonstrated promising results in multiple studies related to brain injury including intraparenchymal hemorrhage, acute stroke, subarachnoid hemorrhage, and general injury to the blood-brain-barrier. 6 hours following intracerebral hemorrhage in adult mice, curcumin was administered in clinically relevant doses of 75-300 mg/kg. After 72 hours, there was a reduction in hematoma size, decreased vasogenic edema secondary to a less damaged blood-brain-barrier, decreased inflammatory markers, and overall improved neurological outcome. After discussing the role of T-lymphocytes in contributing inflammation and worsening neuronal injury, mouse models were used to demonstrate a suppression of T-lymphocyte infiltration in the brain after administration of curcumin. There was also a reduction in cerebral edema and improvement of neurological scores. One study administered low dose (80mg/day) curcumin to healthy middle-aged adults (40-60 years of age), when compared to a placebo group. The CC group had lower levels of plasma triglyceride, salivary amylase levels, plasma beta amyloid protein concentrations (protein responsible for Alzheimer's disease and other forms of intracerebral hemorrhage), and other beneficial health effects.

It was recently detected that combining CC with piperine (black pepper extract, also known as peperine or BioPerine), a known inhibitor of hepatic and intestinal glucuronidation, enhances the serum concentration, extent of absorption and bioavailability of CC in both rats and humans. Therefore, CC supplement is now used in combination with the black pepper extract. The average amount of pepper consumed by a person during a day in the United States is 359 mg, which translates to 18-32 mg of piperine a day. Furthermore, rat trials show a daily intake of 5 to 20 times the average daily dose of humans produced no clinical symptoms. Studies on acute, subacute, and chronic piperine toxicity show no abnormalities or clinical symptomatology, or significant blood chemistry data in laboratory animals. Black pepper extract has a high degree of safety being used nutritionally. The amount of piperine that is formulated in the curcumin capsules is several thousand times less than the LD50 (lethal dose 50) established in mice and rats. Our capsule contains 270 mg of pure curcuminoids (curcumin) and 3mg of black pepper extract. The recommended serving size is 3 capsules a day. Therefore, the patients will receive 810mg of pure curcumin and 9mg of black pepper extract (peperine) per day, which is less than the average amount of pepper consumed by a person daily in the United States.

This is a double-blinded, randomized placebo-controlled pilot study. A total of 48 subjects will be recruited in this study. 24 patients will receive placebo pills, and 24 will receive Curcumin (CC) pills. Patients who have symptomatic unilateral chronic subdural hematomas, with no acute component and do not meet the exclusion criteria, will be evaluated. At the time of consent for evacuation of the subdural hematoma, patients will also be consented for this trial by the research team. Participants will be instructed that they will be randomized to either the placebo group or the curcumin group. Participants will take one capsule three times a day for a maximum of 60 days. Participants will undergo standard postoperative care in regard to imaging and clinical follow-up. Patients will begin taking placebo or CC within 24 hours post-operatively and able to take oral medication. It will then be continued three times a day (TID).

This is a single center study that will take place at the University of New Mexico Hospital (UNMH). New patients admitted directly to the UNM Neurosciences Intensive Care Unit (NSICU) as a transfer from an outside hospital as well as patients admitted directly through the UNM (University of New Mexico) Emergency Department (ED), with subdural hematomas will be identified and recruited as potential subjects. All surgical operations will take place in the main operating room (OR) at UNMH. The perioperative care of the enrolled patients, as well as the non-surgically managed patients will take place both in the NSICU as well as the Neurosurgical step-down unit. Once patients have been discharged from the hospital, all follow-up appointments will take place in the Clinical Neurosciences Center located adjacent to UNMH. Patients will follow-up in the subdural clinic, staffed by Dr. Howard Yonas, Principal Investigator.

ELIGIBILITY:
Inclusion Criteria:

1. Chronic subdural hematoma (cSDH)
2. Age of 18 years old or older
3. Unilateral cSDH with no other intracranial injuries

   o Membranes with minimal hemorrhage may be included but no clear acute component should be evident
4. Subdural volume less than 115cc
5. MARWALDER GRADING SCALE Score of 0-2
6. Patient or patient's power of attorney (POA) is available to sign consent
7. Patient undergoes surgical evacuation of cSDH-

Exclusion Criteria:

1. Age less than 18 years old
2. Bilateral subdural hematomas
3. Subdural volume less than 115cc
4. Acute subdural hematoma
5. Patient does not undergo surgical evacuation
6. Other evidence of intracranial injury (i.e. epidural hematoma, intraparenchymal hemorrhage, skull fractures, subarachnoid hemorrhage, hydrocephalus)
7. Patient's family not available for consent and requires emergent surgical evacuation
8. Previous intracranial surgery
9. Recent head trauma (less than1 week)
10. Use of anti-coagulation (i.e. Coumadin, Heparin, Apixaban, and Rivaroxaban) or antiplatelets (Plavix) drugs, with the exception of Aspirin
11. Known coagulopathy disorders
12. Positive urine or serum pregnancy test in pre-menopausal female subjects, without a documented history of surgical sterilization; or currently breastfeeding (Since the nuclear group in an older population, the pregnancy test will be made in exceptional cases).
13. Allergy to curcumin or turmeric.
14. Allergy to black pepper
15. Markwalder Grading Scale Score: 3-4
16. Baseline dementia (for more than 6 months). Adult who cognitively impaired for more than 6 months will be excluded from the study, since this impairment might be due to other reasons than cSDH, such as dementia or cognitive impairment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2018-12-18 (Actual); Primary Completion 2020-02-26 (Actual); Study Completion 2020-02-26 (Actual)

PRIMARY OUTCOMES:
Measurements by CT of subdural hematoma volume change | 6 months
  Change of the total hematoma cavity volume compared to post-subdural drain removal to volumes of less than 80 cc in post-surgical patients

SECONDARY OUTCOMES:
Recurrence rate of cSDH with and without CC treatment | 6 months
  Change re-accumulation rate of cSDH

OTHER OUTCOMES:
Patient's neurological status | 6 months
  Change rate of persistent or recurrent neurological symptoms

CONTACTS AND LOCATIONS:
Overall Officials: Howard Yonas, MD, Principal Investigator — UNM
Locations (1):
- University of New Mexico Health Sciences center, Albuquerque, New Mexico, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Arbiser JL, Klauber N, Rohan R, van Leeuwen R, Huang MT, Fisher C, Flynn E, Byers HR. Curcumin is an in vivo inhibitor of angiogenesis. Mol Med. 1998 Jun;4(6):376-83. PMID 10780880
- [Background] Asher GN, Spelman K. Clinical utility of curcumin extract. Altern Ther Health Med. 2013 Mar-Apr;19(2):20-2. PMID 23594449
- [Background] Bhandarkar SS, Arbiser JL. Curcumin as an inhibitor of angiogenesis. Adv Exp Med Biol. 2007;595:185-95. doi: 10.1007/978-0-387-46401-5_7. PMID 17569211
- [Background] Brokinkel B, Ewelt C, Holling M, Hesselmann V, Heindel WL, Stummer W, Fischer BR. Routine postoperative CT-scans after burr hole trepanation for chronic subdural hematoma - better before or after drainage removal? Turk Neurosurg. 2013;23(4):458-63. doi: 10.5137/1019-5149.JTN.7269-12.0. PMID 24101264
- [Background] DiSilvestro RA, Joseph E, Zhao S, Bomser J. Diverse effects of a low dose supplement of lipidated curcumin in healthy middle aged people. Nutr J. 2012 Sep 26;11:79. doi: 10.1186/1475-2891-11-79. PMID 23013352
- [Background] Fan X, Zhang C, Liu DB, Yan J, Liang HP. The clinical applications of curcumin: current state and the future. Curr Pharm Des. 2013;19(11):2011-31. PMID 23116310
- [Background] Frati A, Salvati M, Mainiero F, Ippoliti F, Rocchi G, Raco A, Caroli E, Cantore G, Delfini R. Inflammation markers and risk factors for recurrence in 35 patients with a posttraumatic chronic subdural hematoma: a prospective study. J Neurosurg. 2004 Jan;100(1):24-32. doi: 10.3171/jns.2004.100.1.0024. PMID 14743908
- [Background] Gelabert-Gonzalez M, Aran-Echabe E. Can recurrence of chronic subdural hematoma be predicted? J Neurol Surg A Cent Eur Neurosurg. 2014 Sep;75(5):407. doi: 10.1055/s-0033-1358613. Epub 2013 Dec 19. No abstract available. PMID 24357072
- [Background] Ghosh S, Banerjee S, Sil PC. The beneficial role of curcumin on inflammation, diabetes and neurodegenerative disease: A recent update. Food Chem Toxicol. 2015 Sep;83:111-24. doi: 10.1016/j.fct.2015.05.022. Epub 2015 Jun 9. PMID 26066364
- [Background] Gupta SC, Patchva S, Aggarwal BB. Therapeutic roles of curcumin: lessons learned from clinical trials. AAPS J. 2013 Jan;15(1):195-218. doi: 10.1208/s12248-012-9432-8. Epub 2012 Nov 10. PMID 23143785
- [Background] Hennig R, Kloster R. Burr hole evacuation of chronic subdural haematomas followed by continuous inflow and outflow irrigation. Acta Neurochir (Wien). 1999;141(2):171-6. doi: 10.1007/s007010050282. PMID 10189499
- [Background] Hickey MA, Zhu C, Medvedeva V, Lerner RP, Patassini S, Franich NR, Maiti P, Frautschy SA, Zeitlin S, Levine MS, Chesselet MF. Improvement of neuropathology and transcriptional deficits in CAG 140 knock-in mice supports a beneficial effect of dietary curcumin in Huntington's disease. Mol Neurodegener. 2012 Apr 4;7:12. doi: 10.1186/1750-1326-7-12. PMID 22475209
- [Background] Hidaka H, Ishiko T, Furuhashi T, Kamohara H, Suzuki S, Miyazaki M, Ikeda O, Mita S, Setoguchi T, Ogawa M. Curcumin inhibits interleukin 8 production and enhances interleukin 8 receptor expression on the cell surface:impact on human pancreatic carcinoma cell growth by autocrine regulation. Cancer. 2002 Sep 15;95(6):1206-14. doi: 10.1002/cncr.10812. PMID 12216086
- [Background] Hong HJ, Kim YJ, Yi HJ, Ko Y, Oh SJ, Kim JM. Role of angiogenic growth factors and inflammatory cytokine on recurrence of chronic subdural hematoma. Surg Neurol. 2009 Feb;71(2):161-5; discussion 165-6. doi: 10.1016/j.surneu.2008.01.023. Epub 2008 Apr 18. PMID 18423527
- [Background] King MD, McCracken DJ, Wade FM, Meiler SE, Alleyne CH Jr, Dhandapani KM. Attenuation of hematoma size and neurological injury with curcumin following intracerebral hemorrhage in mice. J Neurosurg. 2011 Jul;115(1):116-23. doi: 10.3171/2011.2.JNS10784. Epub 2011 Mar 18. PMID 21417704
- [Background] Lao CD, Ruffin MT 4th, Normolle D, Heath DD, Murray SI, Bailey JM, Boggs ME, Crowell J, Rock CL, Brenner DE. Dose escalation of a curcuminoid formulation. BMC Complement Altern Med. 2006 Mar 17;6:10. doi: 10.1186/1472-6882-6-10. PMID 16545122
- [Background] Lin CC, Lu YM, Chen TH, Wang SP, Hsiao SH, Lin MS. Quantitative assessment of post-operative recurrence of chronic subdural haematoma using mean haematoma density. Brain Inj. 2014;28(8):1082-6. doi: 10.3109/02699052.2014.901559. Epub 2014 Apr 4. PMID 24701968
- [Background] Liu W, Yuan J, Zhu H, Zhang X, Li L, Liao X, Wen Z, Chen Y, Feng H, Lin J. Curcumin reduces brain-infiltrating T lymphocytes after intracerebral hemorrhage in mice. Neurosci Lett. 2016 May 4;620:74-82. doi: 10.1016/j.neulet.2016.03.047. Epub 2016 Mar 26. PMID 27026486
- [Result] Gururaj AE, Belakavadi M, Venkatesh DA, Marme D, Salimath BP. Molecular mechanisms of anti-angiogenic effect of curcumin. Biochem Biophys Res Commun. 2002 Oct 4;297(4):934-42. doi: 10.1016/s0006-291x(02)02306-9. PMID 12359244

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2018-08-29): https://cdn.clinicaltrials.gov/large-docs/22/NCT03845322/Prot_SAP_000.pdf
  • Informed Consent Form (2018-08-29): https://cdn.clinicaltrials.gov/large-docs/22/NCT03845322/ICF_001.pdf